CLINICAL TRIAL: NCT00014352
Title: Phase II Trial Of Sequential Estramustine/Paclitaxel Followed By Doxorubicin/Ketoconazole In Patients With Androgen-Independent Prostate Cancer
Brief Title: Combination Chemotherapy Plus Warfarin in Treating Patients With Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 00-113; MSKCC-00113; NCI-G01-1927
Record Dates: First submitted 2001-04-10; First posted 2003-11-13 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Prostate Cancer; Thromboembolism
Keywords: stage III prostate cancer; stage IV prostate cancer; recurrent prostate cancer; thromboembolism
MeSH Terms: conditions — Prostatic Neoplasms; Thromboembolism | interventions — Docetaxel; Doxorubicin; Estramustine; Ketoconazole; Warfarin

INTERVENTIONS:
Drug: docetaxel
Drug: doxorubicin hydrochloride
Drug: estramustine phosphate sodium
Drug: ketoconazole
Drug: warfarin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. Anticoagulant drugs such as warfarin may reduce the risk of blood clots.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy plus warfarin in treating patients who have prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the safety, efficacy, and durability of docetaxel and estramustine followed by doxorubicin and ketoconazole in patients with high-risk, androgen-independent prostate cancer. II. Determine whether anticoagulation with warfarin can reduce the frequency of thromboembolic complications associated with estramustine in these patients.

OUTLINE: Regimen A: Patients receive oral estramustine 3 times daily on days 1-5 and docetaxel IV over 1 hour on day 3 weekly. Patients also receive oral warfarin daily. Treatment repeats every 4 weeks for a total of 2 courses in the absence of disease progression or unacceptable toxicity. Regimen B: After completion of regimen A, patients receive doxorubicin IV over 30 minutes weekly and oral ketoconazole twice daily. Treatment repeats every 4 weeks for a total of 2 courses in the absence of disease progression or unacceptable toxicity. Patients are followed monthly until disease progression.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed prostate cancer High risk as defined by any 2 of the following: Karnofsky performance status of 70-80% Lactate dehydrogenase greater than 200 U/mL Hemoglobin less than 13 g/dL Prostate-specific antigen (PSA) at least 4 ng/mL Progressive disease based on any 1 of the following: Rise in PSA level of at least 25% above baseline At least 3 determinations taken at weekly intervals OR At least 2 determinations taken at monthly intervals New or progressive soft tissue masses on MRI or CT scan Radionucleotide bone scan with new metastatic lesion(s) Serum testosterone no greater than 30 ng/mL If no prior surgical orchiectomy, castrate levels of serum testosterone must be maintained with continuation of gonadotropin releasing hormone analogs If receiving an anti-androgen, must show progression of disease after stopping anti-androgen therapy

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: See Disease Characteristics Karnofsky 70-100% Life expectancy: Not specified Hematopoietic: See Disease Characteristics WBC at least 3,000/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin normal SGOT/SGPT no greater than 1.5 times upper limit of normal (ULN) Renal: Creatinine no greater than 1.5 times ULN Cardiovascular: No significant cardiovascular disease No New York Heart Association class III or IV heart disease No active angina pectoris No myocardial infarction within the last 6 months Ejection fraction at least 45% by echocardiogram or MUGA No prior hemorrhagic or thrombotic cerebral vascular accident No deep venous thrombosis Pulmonary: No pulmonary embolism within the past 6 months Other: No history of bleeding disorder or gastrointestinal bleeding that would preclude anticoagulation with warfarin No other concurrent malignancy except non-melanoma skin cancer or any curatively treated malignancy considered to be at less than 30% risk of relapse No severe infection No severe malnutrition No other serious medical illness that would preclude study

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No more than 1 prior chemotherapy regimen Endocrine therapy: See Disease Characteristics Radiotherapy: No more than 1 prior course of palliative radiotherapy No more than 1 prior radioisotope therapy with strontium chloride Sr 89 or samarium Sm 153 lexidronam pentasodium Surgery: See Disease Characteristics At least 4 weeks since prior major surgery

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-09; Primary Completion 2003-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William K. Kelly, DO, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States